CLINICAL TRIAL: NCT06593444
Title: The Efficacy and Safety of Thalamic Ventral Intermediate Electrical Stimulation for Refractory Familial Cortical Myoclonus with Epilepsy: a Prospective, Pilot Trial
Brief Title: Thalamic Ventral Intermediate Electrical Stimulation for Refractory Familial Cortical Myoclonus with Epilepsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-213-003
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Epilepsy (treatment Refractory)
Keywords: Deep Brain Stimulation; Thalamic Ventral Intermediate; Refractory Familial Cortical Myoclonus with Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thalamic Ventral Intermediate-DBS group (Experimental): Participants will undergo Thalamic Ventral Intermediate-DBS ON with the individual stimulation parameters determined in the parameter determination period, then continue to receive stimulation for the remainder of the study.
  Interventions: Procedure: Thalamic Ventral Intermediate-DBS

INTERVENTIONS:
Procedure: Thalamic Ventral Intermediate-DBS — Participants will undergo Thalamic Ventral Intermediate-DBS ON with the individual stimulation parameters determined in the parameter determination period, then continue to receive stimulation for the remainder of the study.

SUMMARY:
The primary objective of this research is to study the efficacy and safety of deep brain stimulation (DBS) of Thalamic Ventral Intermediate as adjunctive therapy for alleviating symptoms in refractory familial cortical myoclonus with epilepsy.

DETAILED DESCRIPTION:
This project aims to include 5 participants, and evaluate the effectiveness and safety of Thalamic Ventral Intermediate electrical stimulation in patients with refractory familial cortical myoclonus with epilepsy through a prospective, interventional, unblinded, single-arm clinical trial. It is expected to provide new therapeutic options for patients with refractory familial cortical myoclonus with epilepsy with alternative treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-70, meeting the diagnostic criteria for Refractory Familial Cortical Myoclonus with Epilepsy (FCMTE), meaning that tremors and/or seizures have not significantly improved despite long-term, stable use of current treatment medications, regardless of gender.
* Tremors and seizures severely impact the patients' work and quality of life.
* Experiencing drug resistance or intolerable adverse reactions to medication.
* After being adequately informed about the nature and risks of the study, willing to provide written informed consent before participating in any study-related procedures.
* Willing to adhere to the relevant trial protocol and regulations, including attending follow-up visits and undergoing related examinations within the specified timeframe.

Exclusion Criteria:

* Patients with FCMTE whose symptoms are essentially controlled after standardized medication and other treatments.
* Presence of structural abnormalities in the VIM (ventral intermediate nucleus).
* Presence of an implanted electrical stimulator (e.g., pacemaker, spinal cord stimulator, repetitive nerve stimulator) or metallic implants in the head (e.g., aneurysm clips, cochlear implants). Note: Vagus nerve stimulation (with stable parameters for at least 3 months) is not an exclusion criterion.
* IQ < 55, severe cognitive impairment that prevents participation in the study.
* Pregnant individuals or those planning to conceive within 2 years.
* Presence of progressive neurological diseases such as brain tumors, arteriovenous malformations, or cavernous hemangiomas.
* Presence of other serious neuropsychiatric disorders such as dementia, severe depression (hospitalized in a psychiatric facility within the past 5 years or any suicidal or self-harming tendencies), schizophrenia, or neurodegenerative diseases. Resolved postictal psychiatric or behavioral abnormalities are not an exclusion criterion.
* Conditions that may increase the risk of seizures during or after surgery (e.g., coagulation disorders) or require long-term oral anticoagulants or antiplatelet drugs.
* Other severe physical illnesses, psychiatric disorders, internal diseases, or severe liver or kidney dysfunction; participation in other clinical trials within the past three months.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Severity of Tremors | Up to 3 months after Thalamic Ventral Intermediate-DBS
  A difference in tremor severity before and after treatment according to the TETRAS scale has been observed.

SECONDARY OUTCOMES:
Seizure Responder Rate | Up to 3 months after Thalamic Ventral Intermediate-DBS
  The proportion of patients with a ≥ 50% reduction from Baseline in seizure frequency.
Life quality evaluation | Up to 3 months after Thalamic Ventral Intermediate-DBS
  Percentage change from baseline in Quality of Life in Epilepsy-31 inventory (QOLIE-31) score. The minimum and maximum values, and whether higher scores mean a better or worse outcome.

OTHER OUTCOMES:
Adverse Events | Up to 3 months after Thalamic Ventral Intermediate-DBS
  Rate of adverse events which were judged to be study-related throughout the study.
Serious Adverse Event | Up to 3 months after Thalamic Ventral Intermediate-DBS
  Rate of serious adverse events which were judged to be study-related throughout the study.
Incidence of Sudden Unexpected Death in Epilepsy (SUDEP) | Up to 3 months after Thalamic Ventral Intermediate-DBS
  The number presented is for Definite and Probable SUDEP. The rate is calculated per 1000 subject years of follow-up.

IPD SHARING:
Plan to Share IPD: No